CLINICAL TRIAL: NCT02711020
Title: Psychological Treatment of Depression in Women With Fibromyalgia: Differential Efficacy and Factors Predictive of Outcome
Brief Title: Psychological Treatment of Depression in Women With Fibromyalgia
Acronym: PCTFORDEPFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Universidad Nacional de Educación a Distancia (Other); University of Hertfordshire (Other); University of Memphis (Other); Arborétum (Unknown)
Responsible Party: Principal Investigator, Dr. Guillem Feixas, Full Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fibro2016; PSI2014-57957-R (Other Grant/Funding Number: Ministry of Economy and Competitiveness (Spanish Government))
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Fibromyalgia; Depressive Symptoms
Keywords: Depressive symptoms; Fibromyalgia; Cognitive Behavioral Therapy; Personal Constructs Therapy; Differential Efficacy
MeSH Terms: conditions — Fibromyalgia; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy delivered in individual format.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Personal Construct Therapy (Experimental): Personal Constructs Therapy delivered in individual format.
  Interventions: Behavioral: Personal Construct Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Patients assigned to this arm will receive a maximum of 18 1-hour sessions of Cognitive Behavioral Therapy following the intervention techniques included in various group therapy manuals for patients with fibromyalgia, plus up to three 1-hour boost sessions between 3 and 5 months after the end of therapy. Techniques are adapted to individual format in the following modules: (1) Psychoeducation, (2) Relaxation, (3) Behavioral Activation, (4) Cognitive Restructuring, (5) Problem solving, (6) Assertiveness Training, and (7) Relapse Prevention.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Personal Construct Therapy — Patients will receive a maximum of 18 1-hour sessions of Personal Constructs Therapy plus up to three 1-hour boost sessions between 3 and 5 months after the end of therapy. The intervention will follow a protocol designed specifically for this project based on the clinical experience of a previous pilot study. It will consist of 4 stages: (1) Analysis of patient's request, goals setting, identification of the main dilemmas, and other personal meanings relevant for self and others' construction; (2) feedback on the assessment results and problem reframing in terms of a "dilemma" and/or other personal meanings; (3) work on the dilemmas and/or other aspects of the self and others' construction; and (4) end of the therapeutic process outlining personal projects and future perspectives.
  Other Names: PCT
  Arms: Personal Construct Therapy

SUMMARY:
The purpose of this study is to perform an efficacy study of Personal Construct Therapy, which focuses on the construction of self and others, for women diagnosed with fibromyalgia who have also comorbid depressive symptoms. To that aim, it will be compared with Cognitive Behavioral Therapy, which is an already well-established treatment in this area.

DETAILED DESCRIPTION:
Fibromyalgia is one of the most demanding health issues nowadays due to the high level of suffering and the deterioration of quality of life it entails. In addition, its high prevalence and the great expenses it implies for social and health care systems are also matter of both public and politic concern.

Previous research has shown that the personal affliction triggered by fibromyalgia is influenced by psychological factors, which have also an effect on the socioeconomic burden of this disease as a consequence. Among these factors, depressive symptoms are highlighted in this study not only because they exacerbate the clinical profile of this type of patients, but also because they decrease their response to treatment, contributing to the chronicity of this disease. In fact, the treatment of depressive symptoms is already one of the therapeutic targets included in the most recommended multicomponent (and multidisciplinary) treatment guidelines for fibromyalgia.

In spite of the growing number of studies supporting the efficacy of psychological therapies for fibromyalgia, many issues need further development. For example, current treatment recommendations for this syndrome suggest that the intervention must be tailored to the psychosocial and functioning profile of patients. However, research is still needed in order to enable the identification of key factors for clinical improvement. Similarly, it is crucial to identify and assess idiosyncratic psychological characteristics that may allow the psychological intervention to be effectively adapted. In addition, an evidence-based description of the mechanisms involved in change at different levels (including psychological and physical ones) has not been developed yet.

The aim of this project is to perform an efficacy study of Personal Construct Therapy (PCT), which focuses on the construction of self and others, for women diagnosed with fibromyalgia who have also comorbid depressive symptoms. It will be compared with Cognitive Behavioral Therapy (CBT), which is a well-established treatment in this area. Both interventions will be performed in individual format. Depressive symptoms will be measured before and after treatments, along with other clinical and wellbeing-related variables. The cognitive indexes derived from the Repertory Grid Technique, such as cognitive conflicts, polarization and self-construction measures, will also be assessed. Moreover, the capacity of all these measures for predicting differential outcomes resulting from both treatments will also be estimated. The relevance of these cognitive indicators for depression and fibromyalgia has already been proven by this research group in previous studies.

It is expected that PCT will be more effective than standard CBT in improving clinical symptoms and wellbeing. Additionally, the identification of patients' cognitive characteristics which may have a differential response to the components of each treatment will allow future adaptation of psychological interventions to the characteristics of patients, which will contribute in turn to the improvement of the existing treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of fibromyalgia in the health care system
* A score above 7 on the Hospital Anxiety and Depression Scales

Exclusion Criteria:

* Bipolar disorders
* Psychotic symptoms
* Substance abuse
* Organic brain dysfunction
* Mental retardation
* Serious suicidal ideation
* Receiving psychological treatment (unless it is suspended at the time of inclusion in the study)
* Inability to communicate in Spanish
* Substantial visual, hearing or cognitive deficits

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Hospital Anxiety and Depression Scale at the end of therapy and 6-month follow-up. | End of Therapy (18-30 weeks) and 6-month follow-up (42-54 weeks)
  To assess change in the severity of depressive symptoms with a self-report instrument.

SECONDARY OUTCOMES:
Change from baseline in the Hamilton-Depression Rating Scale at the end of therapy and 6-month follow-up. | End of Therapy (18-30 weeks) and 6-month follow-up (42-54 weeks)
  To assess change in the severity of depressive symptoms with a clinician-administered instrument.
Change from baseline in the Fibromyalgia Impact Questionnaire at the end of therapy and 6-month follow-up. | End of Therapy (18-30 weeks) and 6-month follow-up (42-54 weeks)
  To assess change in the impact of fibromyalgia on functional capacity and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Feixas, Ph.D., Principal Investigator — University of Barcelona
Locations (4):
- Spain (4):
  - Centro de Atención Primaria Les Hortes, Barcelona
  - Centro de Atención Primaria La Guineueta, Barcelona
  - Centro de Salud Mental de Nou Barris Nord, Barcelona
  - Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Paz C, Aguilera M, Salla M, Compan V, Medina JC, Bados A, Garcia-Grau E, Castel A, Canete Crespillo J, Montesano A, Medeiros-Ferreira L, Feixas G. Personal Construct Therapy vs Cognitive Behavioral Therapy in the Treatment of Depression in Women with Fibromyalgia: Study Protocol for a Multicenter Randomized Controlled Trial. Neuropsychiatr Dis Treat. 2020 Jan 24;16:301-311. doi: 10.2147/NDT.S235161. eCollection 2020. PMID 32021219